CLINICAL TRIAL: NCT00936572
Title: A Randomized Double-Blind Trial of Perioperative Administration of Probiotics in Colorectal Cancer Patients.
Brief Title: Probiotics In Colorectal Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02.06.CLI
Record Dates: First submitted 2009-07-07; First posted 2009-07-10 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Colorectal Cancer
Keywords: Probiotics; La1; BB536; Colorectal surgery; Intestinal immunity; Dendritic cells; Lymphocyte; Microbiota
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- high dose (Experimental): high dose of probiotics (109 cfu)
  Interventions: Procedure: Probiotics (La1, BB536)
- low dose (Experimental): low dose of probiotics (107 cfu)
  Interventions: Biological: probiotics (La1, BB536)
- probiotics (Placebo Comparator): Maltodoxtrin
  Interventions: Biological: placebo

INTERVENTIONS:
Procedure: Probiotics (La1, BB536)
  Arms: high dose
Biological: probiotics (La1, BB536)
  Arms: low dose
Biological: placebo — Maltodoxtrin
  Arms: probiotics

SUMMARY:
Design: double blind controlled randomized trial with a parallel design and 3 treatment groups Description of subjects: Patients admitted in study centers for colorectal surgery under laporoscopy and/or laparotomy.

Product:

Product 1: BB536 and LA1 (10E9) Product 2: BB536 and LA1 (10E7) Placebo: Maltodextrin Number of patients: enrolled subjects: n=33, ITT data set: n=31, PP data set: n=30

Primary objective:

Colonization (biopsy+stools) of each bacteria for one of the dose at D0 (surgical procedure)

Secondary objectives:

* Influence of the probiotic bacteria on the gut microflora
* Modulation of the immune and inflammatory response

Additional objectives:

* Investigate dose effect on La1 colonization
* Investigate the effect of La1 colonization, treatment without La1 colonization, and absence of treatment and La1 colonization on other bacteria and on immunological parameters

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

The administration of probiotic bacteria has been hypothesized to affect the composition of the intestinal microflora with reduction of pathogens in favour of non-pathogens. These events might modulate the immune and inflammatory responses, and the gut function.

Experimental data demonstrated that the modulation of the mucosal function and enteric microflora by Lactobacillus plantarum reduces septic morbidity and mortality in animals. The administration of a mix of probiotics has been shown to be more effective than antibiotics to cure pouchitis in humans.

Since patients undergoing colorectal operations have a high risk to develop infections due to the intraoperative contamination with enteral content and the occurence of bacterial translocation, changing the intestinal microflora, by giving lactobacilli may result in important advantages to reduce the risk of intraoperative complications and post operative sepsis.

OBJECTIVES OF THE STUDY

To evaluate if preoperative administration of mucosa reconditioning by probiotic may result in adherence to the colonic mucosa and change of the gut microflora, and may modulate the immune and inflammatory responses and gut function.

EXPERIMENTAL DESIGN AND METHODS

Overall Design and Control Methods Prospective, randomized, double-blind study design.

Centers Departement of Surgery, San Raffaele University, Milan, Italy Departement of Surgery, San Gerardo Hospital, University of Milano-Bicocca, Italy

Number of Subjects/assignment to Formula Groups In these departements about 50 patients are operated for colorectal disease yearly with laparoscopic approach. All these patients are potential candidates to partecipate in the study. It is expected that at least 80% of the patients will agree with partecipation, while during the course of the study about 25% of the partecipants are expected to withdraw. During the intake procedure the inclusion and exclusion criteria are checked. Eligible patients are informed about the objectives, the background and the design of the study. When the patient has given his or her consent to partecipate in the study, the preoperative status is assessed. The patients are then included in the study population and randomly assigned to one of the treatments. During surgery the intraoperative exclusion criteria are checked and non eligible patients excluded from further study. Each group consist of 15 patients in order to assure that at the end of the study 10 patients per group will have completed the study.

Groups:

A: high dose of probiotics (active) compared with B: low dose of probiotics (control) and C: vehicle (placebo)

Dosing Regimen ??

Dosing Scheme:

Preoperative day 5 through 1. Postoperative day 3 through 8. The three preparation will be give 3 times per day (6 hours interval).

Duration of the study 6 months

SCHEDULE OF ASSESSMENTS

Day -6 -1 0 1 2 3 4 5 6 7 8

S

I I I I I MB MB MB MB MB GF GF GF GF GF GF GF GF GF GF

S = select and inform patients I = immunological- inflammatory data MB = microbiological data GF= gastrointestinal function, fecal pH.

Immunological- inflammatory data:

DHR, lymphocyte subset (CD3, CD4, CD8, NK), IgA serum levels, CRP, IL-6, lactate.

Number and subset of intestinal lymphocytes. In vitro response of lymphocytes and macropahges to mitogens and LPS.

Microbiological data:

Quantitative and qualitative culture of stool and colonic mucosa (aerobic and anaerobic total count, aerobic gram negative and positive count)

• During surgery two mucosal samples will be collected for microscopic (adherence test) and microbiological evaluation of the presence of probiotic on the mucosa. Moreover, lymph nodes of the mesentery will harvested for microbiological analysis to assess translocation.

Intraoperative parameters:

Duration of surgery, blood loss, transfusion (amount and type), abdominal contamination.

Gastrointestinal function:

Clinical observation related to gastrointestinal symptoms and defecation pattern

Concomitant Medication and Treatments All patients will receive an antibiotic prophylaxis with cefotetan 2gr 30 minutes before surgery (single shot) and bowel preparation with iso osmotic solution and enema the day before surgery.

STUDY PARAMETERS

Efficacy

Primary Efficacy Parameters

* morphological and microbiological evaluation of the colonic microflora
* gastrointestinal function

Secondary Efficacy Parameters

* immune and inflammatory response
* bacterial translocation

Adverse event

All adverse events encountered during the study will be reported on the Case Report Form. An adverse event is any adverse change from baseline, including intercurrent illness, wich occurs during the course of the study after treatment has started, whether considered related to treatment or not.

Blinding and Randomization

The three study formulae are blinded towards each other. Both researches and patients will be blinded.

Randomization of patients into three groups is performed with the computer randomization program "Random". In this way patient numbers are assigned at random to the group "active formula", "placebo fromula" or "control formula.

Within the three groups randomization is done in blocks of 10 patientnumbers. Per study group three letters are used which are assigned at random to the patientnumbers.

The randomization list may be broken by them in case of an adverse event.

Formulation and Packaging

The formulation of the trial formulae will be in sachet

Dispensing

The investigator is responsible for storage of the study formulae during the time of the study. The sachets must be stored refrigerated until the time of handout. During the actual time that the patient takes the study formula no refrigeration of sachets is required. The investigator is responsible for the hand out of the study formulae in the order of the patientnumber.

A dispensary record of the study formula issued and of any material returned will be kept.

Preparation, Administration and Dosage of test formulae

Route

Before and after the operation the supplement is consumed orally.

Administration protocol For 5 preoperative days in addition of a free choice of hospital food, and after surgery from day 3 to 8.

Assessment of Compliance

The investigator will take high care that patients comply with the conditions set for the study, in order to prevent unnecessary withdrawal because of non compliance.

WITHDRAWAL OF SUBJECTS FROM STUDY

Subjects have the right to withdraw from the study at any time for any reason. The investigator also has the right to withdraw subjects from the study in the event of intercurrent illness, adverse events, treatment failure after a prescribed procedure, protocols violation, cure, administrative reasons or other reasons. It is understood by all concerned that an excessive rate of withdrawal can render the study uninterpretable: therefore, unnecessary, withdrawal of subjects should be avoided. Should subjects decide to withdraw, all efforts will be made to complete and report the observation as thoroughly as possible. A complete final evaluation at the time of the patient's withdrawal should be made with an explanation of why the subjects was withdrawn from the study.

If the reason for removal of a patient from the study is an adverse event or an abnormal laboratory test results, the principal specific event or test will also be recorded on the Case Report Form. In the event of an emergency when the patient's condition requires knowledge of the test treatment, the label may be opened to determine the nature of the test formula dispensed. ANY BROKEN CODE WILL BE CLEARLY JUSTIFIED AND EXPLAINED BY A COMMENT ON THE CASE REPORT FORM, along with the data on which the code was broken.

REPLACEMENT POLICY

Patients withdraw from the study will be replaced if necessary.

CRITERIA FOR EXCLUSION OF SUBJECTS' DATA FROM ANALYSES OF STUDY PARAMETERS

* Intra operative exclusion
* Extensive evidence of non compliance.

Hypothesis Testing

H0: Probiotic bacteria do not affect the microbiology of the gut mucosa and stools gastrointestinal function, immunological or inflammatory parameters compared with control or placebo.

H1: Probiotic bacteria significantly diminishes the number of adhrent and stool pathogens improves gastrointestinal function and/or immunological parameters and/or inflammatory parameters compared with control or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 80 years of age
* Documented cancer disease of the colorectum as diagnos pre-operatively by positive histology.
* Documented bowel disease (IBD, diverticular disease etc) as diagnosed by barium X-Ray or endoscopy.
* Elective colorectal surgery
* Surgical hospital length of stay anticipated to be at least 8 days
* Stool sample available at Day-3 pre-operatively
* Receiving full enteral / oral nutrition
* Written informed consent (by subject or legal guardian)

Exclusion Criteria:

* Perioperative unresectable tumours
* Perioperative neoplastic ascitis
* Emergency colorectal surgery
* Clinically relevant pulmonary or cardiovascular failure
* Liver failure (known cirrhosis or total bilirubin >3 mg/dl)
* Kidney failure (receiving renal dialysis or serum creatinine >2 mg/dl)
* Patients receiving total parenteral nutrition (TPN)
* Immunological disorders
* Ongoing or recent infections (within last 10 days)
* Pregnant (patient's declaration)
* Participation in another clinical trial

SUBJECT SELECTION CRITERIA

* Population Base: Patients with diagnosis of disease of the colorectum, elective for colorectal surgery

Inclusion Criteria:

* Both sexes with age greater than 18 years.
* Documented disease of the colorectum, candidate to major elective surgery.
* Provided written informed consent.

Exclusion Criteria

* Preoperative:

  * clinically relevant failure of the pulmonary
  * cardiovascular, renal or hepatic system
  * ongoing bleeding
  * immunological disorder
  * ongoing or recent infections
  * emergency surgery
* Intraoperative:

  * unresectable tumors
  * neoplastic ascitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Parameters: morphological and microbiological evaluation of the colonic microflora, gastrointestinal function

SECONDARY OUTCOMES:
Secondary Efficacy Parameters: immune and inflammatory response, bacterial translocation

CONTACTS AND LOCATIONS:
Locations (1):
- Gianotti Luca Vittorio, Monza, Italy